CLINICAL TRIAL: NCT05045209
Title: Virtual Exercise Rehabilitation Treatment Program for Post Exacerbation of Chronic Obstructive Pulmonary Disease
Acronym: VERTEX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Natya Raghavan, Principal Investigator, St. Joseph's Healthcare Hamilton
Other Study IDs: 13451
Record Dates: First submitted 2021-09-05; First posted 2021-09-16 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Telerehabilitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Virtual rehabilitation: Virtual pulmonary rehabilitation will be provided by a tablet with connection to a physiotherapist for monitored exercise sessions with educational videos provided on the tablet.
  Interventions: Other: Virtual rehabilitation

INTERVENTIONS:
Other: Virtual rehabilitation — Patient who are assigned to this group will receive virtual rehabilitation

SUMMARY:
Respiratory rehabilitation is an intervention proven to improve quality of life in those with chronic lung disease but access remains poor. The investigators will assess the feasibility and acceptability of a virtual platform for respiratory rehabilitation as an alternative to in person rehabilitation. The aim is to use the technology in those post admission with COPD where access has been even more of a challenge as during this period patients find it difficult to access an out patient program due to their frailty.

DETAILED DESCRIPTION:
People living with lung disease struggle with activities. An exercise program can help but these programs are limited and are hard to get to and generally have a long wait list. The investigators will offer exercise and education through a tablet with internet provided 2 times per week for 10 weeks for patients admitted to hospital with a worsening of their COPD. Patients will work with a trained therapist for the exercise sessions and with the team for the education sessions. The investigators will assess outcomes on functional and quality of life improvements as well as feasibility and scalability of the technology.

ELIGIBILITY:
Inclusion Criteria:

* minimum age of 18 years
* maximum age of 90 years
* diagnosis of COPD

Exclusion Criteria:

* inability to perform exercise
* severe debilitating conditions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admitted patients >40years of age with documented diagnosis of COPD
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test distance | 1 year
  The distance walked during the 6 minute
1-MSTST | 1 year
  One-minute sit to stand test

OTHER OUTCOMES:
Daily activity levels | 1 year
  Measured by step counts

CONTACTS AND LOCATIONS:
Locations (1):
- St. Josephs' Hospital, Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No